CLINICAL TRIAL: NCT00367627
Title: Relative Efficacy of Two Regimens of Ante-helminthic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-026
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2006-08

CONDITIONS: Helminthiasis
Keywords: Children; Malnutrition; Ascaris Lumbricoides; Trichuris trichiura Morbidity; Helminthiasis; Children 2-5 years; Stool RME +ve for helminthiasis
MeSH Terms: conditions — Helminthiasis; Malnutrition | interventions — Albendazole

INTERVENTIONS:
Drug: Albendazole

SUMMARY:
The most common soil transmitted helminthic infections(STHI) includes infection with Ascaris lumbricoides, Trichuris trichiura, and Hookworm. Growth retardation, malnutrition, anemia, impaired cognitive function and immunosuppression are main manifestations in children. Even within the developing world, wide differences exist in prevalence rates. The poorest countries have higher levels of STHI than those with a lower incidence of poverty. According to an estimate made by the WHO, the prevalence of A. lumbricoides, T. trichiura and Hookworm in South Asia was 27%, 20% and 16% respectively. Given that the prevalence of STHI in urban slums in Bangladesh is much higher than the other parts of the world and Asia and that there are major health and socio-economic consequences of such infections, it is important that we come up with effective means of reducing the prevalence of such infections. 60-80% of preschool children in urban slums of Bangladesh are infected with these STHI due to poor hygiene . At present deworming at six months interval is recommended but the effectiveness of this regimen of dewormig is questionable.

2. Hypothesis: Ante-helminthic treatment at every three month is more effective than ante-helminthic treatment at every six months to reduce soil transmitted helminthic infection, to reduce diarrheal and respiratory illness to improve nutritional status in preschool children.

3.Objective: The main objectives of the proposed study is to compare the relative efficacy of two different ante-helminthic treatment regimens to reduce the prevalence of STHI, diarrheal diseases, respiratory illness and to improve nutritional status in children 4. Design: The population of the study will be preschool children aged 2-5 year and will be selected randomly from an urban of Dhaka. They will be divided into two groups randomly. One group will get ante-helminthic at every three months interval and the other groups will get at six months interval for one year. Stool samples will be collected at the baseline and after three months completing one-year treatment of the above mentioned regimen. Blood haemoglobulin and nutritional status will also be measured at baseline and after three months of completion of treatment as mentioned above. The treatment will be 400 mg of Albendazole in a single dose.

5. Potential Impact: The findings of the research can be implemented by the government and non-government organization.

DETAILED DESCRIPTION:
Study design and population:

The study population will be the children aged 2-5 years old in the study area. All children aged 2-5 years old in one slums of the study area will be listed and will be invited to participate in the study.

Parents will be explained the purpose of the study and will be asked for written consent for participation of their children in the study. If the parents give the consent then a stool pot will be given to them to collect stool samples for microscopic examination for intestinal parasites. The inclusion criteria are; 1) age of the child is 2-5 years old, 2) he/she has not been suffering from serious chronic illness, 3) the child stool test must be positive for STH, 4) he/she had not been taken any antehelminthic drug in the previous six months, 5) parents/guardian are agree for their child participation in the study. The exclusion criteria are; 1) age of the child less than 2 years old and more than 5 years old, 2) his/her stool test negative for any intestinal helminth, 3) he/she has been suffering from serious chronic illness, 4) parents/guardian are not willing to give consent for their child's participation in the study, 5) if he/she receives any antehelminthic drug after survey but before the study interventions. The survey will be done in the first months of the study, and then children will be enrolled according to above mentioned inclusion/exclusion criteria. During screening if any child is found severely malnourished it will be considered as'danger sign' according to WHO and IMCI guideline he/she will be referred to an appropriate facility even if she/he is not enrolled in the study. Simple randomization technique will be applied to divide the children into two groups: A) Conventional treatment group who will receive anti-helminthic treatment 400 mg of Albendazole in a single dose at six month interval and B) Intervention group, who will receive anti-helminthic 400 mg of Albendazole in a single dose treatment at three months interval. Stool samples will be collected from both groups prior to anti-helminthic therapy and will be examined quantitatively. However stool examination will not be carried out for intestinal parasite after giving 400 mg of Albendazole at 12 months.

Sample size calculation:

Sample size has been calculated using different predicted values of different out come variables and is shown in the Table 1. A sample size of 200 children, 100 in each group will be sufficient for the study.

Table 1. Sample size calculation table Indicator Conventional treatment group Intervention treatment group Power of the study 95% CI SD* Number in each group Total number adjusted for 10% drop out Cure rate 40% 65% 90% 95% - 78 170 HAZ < -2 38% 19% 90% 95% - 84 184 Incidence of E. histolytica infection per 100 child-year 20a 15 90% 95% 10 85 188 Average diarrheal episode per child 2a 1 90% 95% 1.5 48 106 Mean haemoglobin mg% 10a 12 90% 95% 4 85 188 Respiratory tract infection episode/child 6a 4 90% 95% 3 48 106 * SD = Within group standard deviation

a= Data from our ongoing cohort study in Mirpur

Methods:

Anthropometric measurement: Field Research Assistant will be trained to take weight and height measurement of the children. Anthropometric measurements will be taken by trained FRA at the time of enrollment and then every 3-months. Each child will be weighed in light clothes with an electronic weighing scale. Inter-observer variation up to 2.5% will be allowed. The standing heights of children will be measured to the nearest 0.1 cm using a locally constructed height stick. Again inter-observer variation up to 2.5% will be allowed. Nutritional status will be assessed by comparing the weight and height of the study children with those of NCHS reference population of the same age and sex with the help of Epi6 computer package program and weight for age "Z" score (WAZ) and height for age "Z" score (HAZ) will be computed (29). Malnourished and stunted will be defined by the WAZ score and HAZ score <-2 respectively.

Other disease morbidity: Each study subject will be visited by a community health worker every week and will collect information by asking parents/guardian according to structured questionnaires about diarrheal disease, fever, cough etc. of the child retrospectively for previous seven days. They will work 6 days weekly and every one of them has to visit about 17 households per day for morbidity data collection. Parents/guardian will be advised to seek health care from study physician in study field office in case of any illness of the study child. The study physician will take history and will carry out physical examination and will give treatment to the sick child. If the child does not respond to the given treatment or if his/her condition deteriorates or if the child is seriously ill initially then he/she will be referred to the appropriate referral facilities for treatment, and treatment cost will not be carried out by the project. Asymptomatic E. histolytica infections will not be treated. But symptomatic E. histolytica infections will be treated according to the ICDDR, B Dhaka Hospital treatment guidelines

Intestinal helminth infections induce Th-2 immune response (27), which might favor others viral, bacterial and protozoan infections. De-worming has been shown to improve antibody response (28). In our ongoing cohort study in Mirpur it has been found that children with heavy Trichuris trichiura (TT) infections suffered significantly more from E. histolytica associated infection (un published data) compare to those children with light infection with TT. Based on these observations it can be hypothesized that a frequent de-worming regimen will be associated with less other disease morbidtity like diarrheal diseases, respiratory infections and intestinal protozoan infections with E. histolytica Clinical definitions Diarrhea was defined as having three or more unformed stools in a 24 hour period. A "diarrheal episode" was defined as being separated from another episode by at least 3 diarrhea-free days.

Respiratory tract infection defined as a 'Perceptions of a child who has a cough, is breathing faster than usual with short, quick breaths or is having difficulty breathing, excluding children that had only a blocked nose. (30). No attempt will be done to identify the etiology of the respiratory infection.

Cure rate of STH infection (CR): Cure rate from STH infection is defined as follows:

* Prevalence before at enrollment - % prevalence at the end of the study CR = --------------------------------------------------------------------------------------------- x 100%
* Prevalence before at enrollment

Laboratory methods:

Blood hemoglobin measurement: Study physician will measure blood hemoglobin of the child at enrollment and at the end of the study period by hemocytometer at field site. (31).

Stool parasite examination: The community health workers will collect stool samples for qualitative and quantitative intestinal parasite measurement at every three months interval. The stool will be examined by conventional microscopy for qualitative measurement and for quantitative measurement of intestinal helminthes by Kato-Katz or Formalin-ether concentration technique will be used. (32).E. histolytica will be detected by stool microscopy and ELISA as described by R Haque el at(33).

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria are;

1. age of the child is 2-5 years old,
2. he/she has not been suffering from serious chronic illness,
3. the child stool test must be positive for STH,
4. he/she had not been taken any antehelminthic drug in the previous six months,
5. parents/guardian are agree for their child participation in the study. e -

Exclusion Criteria:

1. age of the child less than 2 years old and more than 5 years old,
2. his/her stool test negative for any intestinal helminth,
3. he/she has been suffering from serious chronic illness,
4. parents/guardian are not willing to give consent for their child's participation in the study,
5. if he/she receives any antehelminthic drug after survey but before the study interventions.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To determine the relative efficacy of de-worming at every three months vs. every six month single dose of Albendazole treatment.

SECONDARY OUTCOMES:
To compare additional morbidity information such as diarrheal diseases, respiratory tract infections, nutritional status and E. histolytica associated morbidity between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad M Alam, MBBS, Principal Investigator — ICDDR,B: Centre for Health and Population Research
Locations (1):
- ICDDR,B: Centre for Health and Population Research, Dhaka, Bangladesh